CLINICAL TRIAL: NCT01645930
Title: A Phase 1 Pharmacokinetic and Tolerability Study of Oral MLN9708 Plus Lenalidomide and Dexamethasone in Adult Asian Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Phase 1 Pharmacokinetic Study of Oral Ixazomib Plus Lenalidomide and Dexamethasone in Adult Asian Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16013; U1111-1155-5943 (Registry Identifier: WHO); HKUCTR-1593 (Registry Identifier: HKUCTR)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ixazomib+Lenalidomide+Dexamethasone (Experimental): Ixazomib 4 mg, capsules, orally, once on Days 1, 8, and 15; lenalidomide 25 mg, capsules, orally, once on Days 1 through 21; and dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15, and 22 of a 28-day treatment cycle until progressive disease (PD) or unacceptable toxicity (up to 20 cycles)
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
Drug: Lenalidomide — Lenalidomide capsules
Drug: Dexamethasone — Dexamethasone tablets

SUMMARY:
The purpose of this Phase 1 study is to characterize the pharmacokinetic (PK) and tolerability of oral ixazomib (MLN9708) when administered in combination with lenalidomide and dexamethasone in adult Asian participants with relapsed and/or refractory multiple myeloma.

DETAILED DESCRIPTION:
The drug being tested in this study was ixazomib. Ixazomib was tested to treat adult Asian people who had relapsed and/or refractory multiple myeloma.

The study enrolled 43 patients. Participants were enrolled to receive:

* Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg.

All participants were asked to take ixazomib capsules orally on Days 1, 8, and 15; lenalidomide capsules, orally, on Days 1 through 21; and dexamethasone tablets, orally, on Days 1, 8, 15, and 22 of a 28-day treatment cycle until progressive disease (PD) or unacceptable toxicity (up to 20 cycles).

This multi-center trial was conducted in Singapore, Hong Kong and South Korea. The overall time to participate in this study was up to 577 days. Participants made multiple visits to the clinic, and were contacted 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female East Asian participants 18 years or older
* Diagnosed Multiple Myeloma according to standard criteria
* Measurable disease as specified in study protocol
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Participants with relapsed and/or refractory Multiple Myeloma who have received 1 to 3 prior therapies
* Meet the clinical laboratories criteria as specified in the protocol
* Female participants who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to abstain from heterosexual intercourse; must also adhere to the guidelines of the lenalidomide pregnancy prevention program
* Male participants who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse and must adhere to the guidelines of the lenalidomide pregnancy prevention program
* Must be able to take concurrent aspirin 325 mg daily
* Voluntary written consent

Exclusion Criteria:

* Female participants who are lactating or pregnant
* Major surgery or radiotherapy within 14 days before enrollment
* Infection requiring systematic antibiotics within 14 days before study enrollment
* Central nervous system involvement
* Failure to have fully recovered from the effects of prior chemotherapy regardless of the interval since last treatment
* Systemic treatment with strong inhibitors of cytochrome P450 1A2 (CYP1A2), strong inhibitors of CYP3A, or strong CYP3A inducers, or use of Ginko biloba or St. John's wort within 14 days before study enrollment
* Diagnosis of Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes) syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome
* Evidence of current uncontrolled cardiovascular conditions
* Serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol
* Known allergy to any of the study medications
* Known gastrointestinal condition or procedure that could interfere with swallowing or the oral absorption of tolerance of ixazomib
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease with the exception of nonmelanoma skin cancer or any completely resected carcinoma in situ
* Ongoing or active systemic infection, active hepatitis B virus infect, active hepatitis C infection, or known human immunodeficiency virus (HIV) positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-12-17 (Actual); Primary Completion 2014-07-14 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (5):
- Hong Kong (2):
  - Pokfulam
  - Shatin
- Singapore, Singapore
- South Korea (2):
  - Incheon
  - Seoul

REFERENCES:
- [Derived] Gupta N, Goh YT, Min CK, Lee JH, Kim K, Wong RS, Chim CS, Hanley MJ, Yang H, Venkatakrishnan K, Hui AM, Esseltine DL, Chng WJ. Pharmacokinetics and safety of ixazomib plus lenalidomide-dexamethasone in Asian patients with relapsed/refractory myeloma: a phase 1 study. J Hematol Oncol. 2015 Sep 4;8:103. doi: 10.1186/s13045-015-0198-1. PMID 26337806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in Singapore, Hong Kong and South Korea from 17 December 2012 to 11 April 2017. Data cut-off for the analysis was 14 July 2014.
Pre-assignment Details: Asian participants with a diagnosis of relapsed and/or refractory multiple myeloma were enrolled and received a combination of ixazomib, lenalidomide and dexamethasone.
Period: Overall Study
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Started | 43
Completed | 0
Not Completed | 43
Not completed — Participants Ongoing on Study Treatment | 22
Not completed — Progressive Disease | 12
Not completed — Adverse Event | 4
Not completed — Unsatisfactory Therapeutic Response | 2
Not completed — Withdrawal by Participant | 2
Not completed — Reason not Defined | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of study drug.
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 43
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 21
  Hong Kong | 6
  Korea, Republic Of | 16
Height at Baseline [Mean (Standard Deviation); unit: cm] | 160.2 (7.80)
Weight at Baseline [Mean (Standard Deviation); unit: kg] | 60.6 (10.47)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Ixazomib
Time Frame: Cycle 1, Day 1 pre-dose and multiple time-points (up to 168 hours) post-dose
Population: Participants from the Pharmacokinetic (PK)-evaluable population, all participants who received protocol-specified dosing during Cycle 1, did not receive any excluded concomitant medications and had sufficient concentration-time data to permit reliable estimation of PK parameters, with data available for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 22
ng/mL | 37.57 (31.701)

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Ixazomib
Time Frame: Cycle 1, Day 15 pre-dose and multiple time-points (up to 336 hours) post-dose
Population: PK-evaluable population included all participants who received protocol-specified dosing during Cycle 1, did not receive any excluded concomitant medications and had sufficient concentration-time data to permit reliable estimation of PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 24
ng/mL | 57.57 (38.507)

3. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Ixazomib
Time Frame: Cycle 1, Day 1 pre-dose and multiple time-points (up to 168 hours) post-dose
Population: Participants from the PK-evaluable population, all participants who received protocol-specified dosing during Cycle 1, did not receive any excluded concomitant medications and had sufficient concentration-time data to permit reliable estimation of PK parameters, with data available for analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 22
hours | 1.5 [0.5 to 7.0]

4. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Ixazomib
Time Frame: Cycle 1, Day 15 pre-dose and multiple time-points (up to 336 hours) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 24
hours | 2.0 [0.5 to 7.97]

5. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for Ixazomib
Time Frame: Cycle 1, Day 1 pre-dose and multiple time-points (up to 168 hours) post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 20
hr*ng/mL | 685.9 (246.35)

6. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration for Ixazomib
Time Frame: Cycle 1, Day 15 pre-dose and multiple time-points (up to 336 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 24
hr*ng/mL | 1746.0 (798.60)

7. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following AEs that were considered by investigator to be possibly related to therapy: 1. Grade 4 neutropenia lasting at least 7 consecutive days; 2. Grade 3 neutropenia with fever and/or infection; 3. Grade 4 thrombocytopenia at least 7 consecutive days; 4. Grade 3 thrombocytopenia with clinically significant bleeding; 5. Platelet count <10,000/mm^3; 6. Grade 2 peripheral neuropathy with pain or ≥Grade 3 peripheral neuropathy; 7. Grade 3 or greater nausea and / or emesis despite the use of optimal anti-emetic prophylaxis; 8. Grade 3 or greater diarrhea that occurred despite maximal supportive therapy; 9. Any other Grade 3 or greater nonhematologic toxicity with the following exceptions: Grade 3 arthralgia/myalgia, <1 week Grade 3 fatigue; 10. A delay of >2 weeks in the subsequent cycle of treatment; 11. Other combination study drug-related nonhematologic toxicities ≥Grade 2 that, in the opinion of the investigator, required discontinuation of study drug.
Time Frame: Cycle 1 (up to Day 28)
Population: DLT-evaluable population consisted of participants who either had a DLT during Cycle 1 or received all scheduled doses and completed all study procedures in Cycle 1 without having a DLT.
Measure: Number; unit: participants
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 24
participants | 2

8. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A SAE is defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or was a medically important event.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 577 days)
Population: Safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 43
participants
  AEs | 43
  SAEs | 18

9. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Reported as Adverse Events of ≥Grade 3 Intensity
Description: Clinically significant laboratory abnormalities were defined as any test results which were observed beyond the clinically acceptable limits as per the discretion of investigator. Clinical laboratory tests included chemistry, hematology and urinalysis tests.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 577 days)
Population: Safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 43
participants
  Alanine Aminotransferase Increased | 2
  Aspartate Aminotransferase Increased | 1
  Blood Creatinine Increased | 1
  Haemoglobin Decreased | 1
  Neutrophil Count Decreased | 2
  Platelet Count Decreased | 4
  Anaemia | 6
  Febrile Neutropenia | 1
  Neutropenia | 12
  Thrombocytopenia | 8
  Hyperglycaemia | 1
  Hypocalcaemia | 3
  Hypokalaemia | 5
  Hypomagnesaemia | 1
  Hyponatraemia | 1
  Hypophosphataemia | 2

10. Primary Outcome: Number of Participants With Clinically Significant Vital Signs Reported as Adverse Events
Description: The number of participants who meet markedly abnormal criteria for vital signs, included diastolic and systolic blood pressure, heart rate, oral temperature, respiratory rate, and body weight.
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug (up to 577 days)
Population: Safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 43
participants
  Grade 1 or 2 Hypertension | 4
  Grade 2 Hypotension | 1

11. Secondary Outcome: Percentage of Participants With Confirmed Best Response Category
Description: Percentage of participants who achieve or maintain any best response category during the treatment period were reported. Best response includes complete response (CR), very good partial response (VGPR), and partial response (PR). Response was assessed according to IMWG criteria. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and ≤5% plasma cells in bone marrow; PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg per 24 hours. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hour.
Time Frame: From Cycle 1, Day 1 to Cycle 3, Day 1 until disease progression (approximately 20 months)
Population: Safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 43
percentage of participants | 53.5

12. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the length of time between the date of first documented response (PR, VGPR, or CR) and the date of first documented progressive disease (PD). According to IMWG criteria: CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and ≤5% plasma cells in bone marrow; PR: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg per 24 hours. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hour.
Time Frame: From date of documentation of a confirmed response to date of progressive disease, (approximately 20 months)
Population: Safety population was defined as all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
Number analyzed (Participants) | 43
months | 12.9 [1.8 to 15.0]

ADVERSE EVENTS:
Time Frame: First dose of study drug through 30 days after the last dose of study drug (up to 577 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ixazomib+Lenalidomide+Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 18/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib+Lenalidomide+Dexamethasone (N=43)
Pneumonia (Infections and infestations) | 3
Lung infection (Infections and infestations) | 2
Diarrhoea infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Gastritis atrophic (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyrexia (General disorders) | 1
General physical health deterioration (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Food allergy (Immune system disorders) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Presyncope (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib+Lenalidomide+Dexamethasone (N=43)
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 12
Cataract (Eye disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 14
Pyrexia (General disorders) | 8
Oedema peripheral (General disorders) | 6
Asthenia (General disorders) | 5
Influenza like illness (General disorders) | 5
Upper respiratory tract infection (Infections and infestations) | 15
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 7
Platelet count decreased (Investigations) | 7
Blood creatinine increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 4
Weight decreased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 12
Hypokalaemia (Metabolism and nutrition disorders) | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 12
Neuropathy peripheral (Nervous system disorders) | 9
Hypoaesthesia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 4
Lethargy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Rash pruritic (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 5
Rash macular (Skin and subcutaneous tissue disorders) | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application